CLINICAL TRIAL: NCT05553379
Title: Clinical Study of the Vivatmo proTM for Fractional Exhaled Nitric Oxide (FeNO) Monitoring in Asthmatic Patients Responding to Inhaled Corticosteroid (ICS) Treatment
Brief Title: Vivatmo proTM EU-study: FeNO Monitoring in Asthmatic Patients Responding to ICS Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bosch Healthcare Solutions GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MDQ-01.736-010-02-EBA-PAM
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Children 7 to 17: Children with asthma
  Interventions: Diagnostic Test: FeNO measurement
- Adults 18 to 80: Adults with asthma
  Interventions: Diagnostic Test: FeNO measurement

INTERVENTIONS:
Diagnostic Test: FeNO measurement — FeNO measurement at each visit

SUMMARY:
This is a multi-center study to evaluate fractional exhaled nitric oxide (FeNO) measured with the Vivatmo pro in adult and pediatric subjects.

DETAILED DESCRIPTION:
Subjects will be screened, enrolled and tested at Study Visit #1 and then prescribed inhaled corticosteroid (ICS) treatment as per routine clinical care. Subjects will return for Study Visit #2 in two weeks and repeat fractional exhaled nitric oxide (FeNO) measured with the Vivatmo pro,

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 7 to 80 years of age.
2. Has asthma
3. Has been identified as a candidate for inhaled corticosteroid (ICS) treatment
4. Is willing and able to perform Vivatmo pro™ testing

Exclusion Criteria:

1. Subject has used corticosteroids prior to enrollment.
2. Subject has other current serious medical conditions
3. Subject has not been clinically stable for at least 2 weeks prior to the study
4. Subject is unwilling or unable to perform Vivatmo pro testing

Ages: 7 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Asthma
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in FeNO Value [Time Frame: 14 days] | 14 days
  Change in FeNO value before and after inhaled corticosteroid treatment

CONTACTS AND LOCATIONS:
Locations (5):
- Czechia (4):
  - MUDr. Ingeborg Vokálova s.r.o, Kralupy nad Vltavou
  - Alergologie Skopkova, s.r.o, Ostrava
  - Plicní středisko Teplice s.r.o, Teplice
  - MUDr. Ivan Drnek, Ústí nad Labem
- Kinderpneumologie und Allergologie im Facharztzentrum, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Registration study for internal use only.